RANDOMIZED CLINICAL TRIAL OF DIATHERMY VERSUS SCALPEL IN ABDOMINAL WALL INCISION DURING REPEAT CESAREAN DELIVERY

Principal Investigator: Martin Caliendo, M.D.

. Martin Canonao, M.B.

Department of Obstetrics and Gynecology, Odessa, TX

Sub-Investigator: Leela Sharath Pillarisetty, M.D, PGY3.

**INTRODUCTION / BACKGROUND** 

Cesarean delivery (CD) is the operative mode of the delivery, which includes laparotomy (skin incision) and hysterotomy (uterine incision) in order to facilitate the delivery of the newborn. In the modern obstetric practice in the United States one in three women who gave birth did so by CD. (1). Cesarean birth can be life-saving for the fetus, the mother, or both in certain cases. The rate of primary CD has increased and more women prefer elective repeat cesarean delivery (ERCD) (2). This increased rate of cesarean deliveries is associated with the short- and long-term maternal complications (3) such as RBC transfusion (2). Among approaches used to reduce the rate of the postoperative complications are prophylactic administration of antibiotics (4) and improvement of surgical techniques (5). In particular, the improvement of surgical technique could contribute to more than two-fold decrease in post-operative morbidity (5). The application of techniques of the abdominal incision during CD is associated with hysterotomy approaches and subsequently maternal morbidity in specific patient populations (6).

During surgical procedures, one of the widely used approaches to decrease blood loss, surgery time and thus post-operative complications is tissue dissection by electrosurgery, which is defined as the process of applying high-frequency electric current to the tissues to cut, coagulate, and desiccate (7). After the introduction of electrosurgery into the practice of surgery in 1926 by William T Bovie and Dr. Harvey W Cushing (8), it has since become a powerful tool in different surgical subspecialties (9)(7).

Protocol version: 1.0 Page **1** of **11** 

Texas Tech University Health Sciences Center IRB NUMBER: L15-144 IRB APPROVAL DATE: 06/17/2015

Electrosurgical instruments are widely used for tissue dissections and to control

bleeding, as an easy and safe surgical approach, but their use in making skin incisions

is limited. The major purported disadvantages of electrosurgical skin incisions are fears

of deep burns; with resultant scaring (10), slower wound healing, and increased

postoperative pain. However, recent meta-analyses showed decreased incision time,

blood loss and post-operative pain with no significant difference in wound infection rates

or scar (13)(14).

With improved techniques of electrosurgery, several randomized trials - the gold

standard of clinical research, were performed. A randomized double blind study (15)

performed in 369 patients, showed that diathermy incision is superior compared to

scalpel incision with reduced incision time, less blood loss and reduced early

postoperative pain. The same advantages have been reported using advanced

diathermy technology by Lee et al(16). The mechanism of these positive effects of

cutting electrosurgey is that the skin is cut with an electrode delivering pure

sinusoidal current, which allows tissue cleavage by rapid cell vaporization without

damage to surrounding areas; this may explain the absence of tissue charring and the

subsequent healing with minimal scarring (17).

Taking together, the recently published advantages of diathermy in the skin incision

could be extremely useful in preventing complications and decreasing maternal

morbidity associated with CD. However, there are no clinical trials comparing scalpel

and diathermy in the population of pregnant patients undergoing CD. To perform such

trials will have direct translational value. In situations of emergency cesarean sections,

as an example, it will provide important information on which method will be fastest with

the least amount of blood loss.

**OBJECTIVE** 

The objective of this study is to compare scalpel vs. diathermy in abdominal wall

incision, in pregnant patients undergoing repeat elective cesarean delivery.

Protocol version: 1.0

**HYPOTHESIS** 

We hypothesize that the abdominal wall incisions made by diathermy compared to

scalpel during repeat cesarean delivery will have less incision time, as well as less

blood loss. Further we hypothesize that the use of diathermy, compared with scalpel will

not increase post-operative pain.

**METHODS** 

1) This is a randomized prospective study in women undergoing elective repeat

cesarean delivery or repeat unplanned non-emergent cesarean delivery at

Medical Center Hospital in Odessa Texas.

2) After informed consent is obtained, women undergoing cesarean delivery will be

randomized into two groups:

Group One

Will undergo diathermy to incise the entire abdominal wall, which includes skin,

subcutaneous tissue, rectus muscle until the peritoneal cavity is visible.

**Group Two** 

Scalpel will be used to achieve the same aims

3) Only patients undergoing elective repeat cesarean delivery will be enrolled, this

will decrease the likelihood of introducing bias into the outcome measures, as

well as it will make the population more uniform.

4) A standardized abdominal wall incision will be made with either diathermy in cut

mode or scalpel. Diathermy will be set in a cut mode with standard setting as per

surgeon's preference. All patients in the study will get standard skin incision in

terms of length and depth which will be marked by a ruler.

5) Incision start and stop time will be recorded by a "timer". A digital wall clock in

the OR will be used to establish time. The timer will instruct the surgeon to "cut".

The timer will record the time. Once the surgeon reaches the abdominal

peritoneum, they will announce "stop". The timers will record the time. The

incision time will be the difference between the "cut" and "stop" times. These

times will be recorded in units of seconds.

Protocol version: 1.0

Texas Tech University Health Sciences Center

6) Along the incision depth the bleeding points will be mopped with sponge laps, no

suction will be used and total blood loss will be calculated by weighing the laps.

7) Blood loss will be recorded as follows: A "used" lap sponge will weighed. A

"fresh" lap sponge will be weighed. These weights will be recorded. Blood loss

will be calculated as the differences in these two weights. These weights will be

recorded in grams.

8) As per standard of care spinal or epidural anesthesia will be administered by

certified registered nurse anesthetist (CRNA). Post-operative pain will be

managed as follows: 1) 300 micrograms of Morphine sulfate will be injected

through then spinal needle or epidural catheter at the beginning of the case. 2)

30 milligrams of Toradol will be injected IM, in the left thigh, at the conclusion of

the case. 3) 10 mg hydrocodone/325mg acetaminophen 1-2 tablets, per oral,

every 4-6 hours, PRN pain.

9) Post-operative pain will be measured by a Numeric Pain Rating Scale (see

below) scored as 0= no pain, up to 10= worst possible pain. This score will be

assessed daily by resident staff at 6:00 to 7:00 AM from post -op day 1 until

hospital discharge.

10) As per standard MCH protocol, within one hour preoperatively, Ancef 2-3 gms will

be administered IV. If the patient is Penicillin allergic, she will receive either 900

milligrams of Clindamycin or 1gram of Vancomycin.

**OUTCOMES-**

Both groups will be assessed for

**Primary outcomes:** 

1. Incision time

2. Blood loss

Secondary outcome:

1. Postoperative pain

Protocol version: 1.0

Texas Tech University Health Sciences Center

SELECTION OF PATIENTS

Inclusion Criteria -

1. Multiparous pregnant women 18 – 45 years.

2. Gestational ages 37 weeks to 41 weeks,

3. Undergoing repeat elective or repeat unplanned non-emergent cesarean

deliveries.

Women with medical comorbidities like hypertension, diabetes complicating

pregnancy, pregnant women with or without prenatal care, and multiple

gestations will also be included.

Exclusion Criteria -

1. Informed consent can't be obtained in a manner that allows for no impression

of undue influence/pressure or sufficient time for patient to consider

participation.

2. Primary Cesarean deliveries – as these can bias the selection.

3. Skin conditions such as infections, psoriasis, and eczema.

**RECRUITMENT PLAN** 

Patients from University Women's Health Centre (Texas Tech OBGYN clinic) and also

from Medical Center Hospital, Odessa, Texas will be recruited. Potential participants will

be identified by a member of the study team or clinic/hospital personnel caring for the

patient. In the latter case, study personnel will be contacted to meet the patient after the

patient has expressed an interest in learning more about participation. All the

participants will have the study procedures, risks, benefits and alternatives explained by

a member of the study team.

Once informed consent is obtained they will be randomized with 1:1 allocation by a

computer generated randomization process. Since the annual rate of cesarean

Protocol version: 1.0

Texas Tech University Health Sciences Center

deliveries in the above-mentioned centers ranges 150 to 175, we expect to enroll a total of 100 patients, and we will allocate 50 patients to each group. Assuming a significance level of 0.05 and a power of 80%, and observing that there is a single measurement and null attrition rate, we will be able to detect at least moderate effect sizes (d=0.50) when performing independent means comparisons.

### **RISKS:**

Diathermy –

- A. Possibility of poor wound healing,
- B. There are concerns that large or excessive scars may form,
- C. Unanticipated burns on skin, subcutaneous tissues and other vital organs.

Scalpel -

- A. Injury to the major blood vessels.
- B. Injury to the vital organs.
- C. Excessive bleeding

From the review of recent literature there are some concerns raised regarding the use of diathermy for skin incisions (10, 11, 12). However, we believe that the use of cutting diathermy, as described in our protocol, does not increase patient risk within the study group. First, there is a concern that diathermy, while making skin incisions, may increase the risk of wound complications, as well as delayed wound healing. However these studies differ from ours in a number of ways: A) Most studies claiming increase in risk examine midline abdominal incisions, and our study employs Pfannenstiel skin incision. B) In some studies it is unclear if pure cut mode was employed. The use of a blend mode will cause more lateral spread of current. This may increase the amount of tissue damage, thus promoting wound complications. Our study will employ diathermy only in pure cut mode in a standard setting as per surgeon's preference. A recent Cochrane review, which includes only randomized trials (the highest form of scientific inquiry), found no significant difference in wound complications between scalpel and diathermy (18).

Protocol version: 1.0

Page **6** of **11** 

Second, there has been a case report of a severe burn injury on patients back while

utilizing diathermy during cesarean delivery (19). The purported mechanism for this

burn was an interaction between diathermy and amniotic fluid (19). However in our

study, cutting diathermy will be used only in incision of skin, subcutaneous fat and

rectus fascia. This use precludes any interaction between diathermy and amniotic fluid.

<u>ADVERSE EVENTS REPORTING:</u>

Any event deemed as an Adverse Event that is possibly related or unexpected to the

study will be assessed at each data gathering point and will be reported to the TTUHSC

IRB as described in the IRB policies and procedure manual. Monitoring of adverse

events will start on the day of surgery.

**BENEFITS** – There are no guarantees of any benefit to study participants. However,

participants may have potential benefits of using electrosurgery which include reducing

the amount of blood loss, dry and rapid separation of tissues. For surgeons, there is a

reduced risk of accidental cut injuries.

**DATA ANALYSIS:** 

Distributions of operative time, blood loss and post-operative pain will be tested for

normal distribution. Student's T test or the non-parametric equivalent will be used to

compare these outcomes between the study and control group. Significance level will

be set at 0.05.

DATA MONITORING PLAN:

All data for each participant will undergo quality assurance monitoring by personnel not

listed as a member of the study team. The purposes of this monitoring are to verify that:

(a) The rights and well-being of human subjects are protected.

(b) The reported trial data are accurate, complete, and verifiable from source

documents.

Texas Tech University Health Sciences Center

Protocol version: 1.0

(c) The conduct of the trial is in compliance with the currently approved protocol/amendment(s), with GCP, and with the applicable regulatory requirement(s).

### **RESULTS**

Expected results will be the finding of less operative time, blood loss, postoperative pain, in diathermy abdominal wall incisions compared to scalpel incisions, in pregnant women undergoing repeat cesarean deliveries.

### **CONCLUSION**

To our knowledge, this study will be the first to compare the results of diathermy vs scalpel abdominal wall incisions in pregnant women undergoing cesarean deliveries.

The study results can be used to help determine which method of incision is preferably used especially in case of emergency cesarean deliveries where time is a crucial factor.

# **Numeric Pain Rating Scale:**



## **REFERENCES-**

1. Obstetric care consensus no. 1: safe prevention of the primary cesarean delivery. Obstetrics and gynecology. 2014;123(3):693-711. Epub 2014/02/21. doi: 10.1097/01.AOG.0000444441.04111.1d. PubMed PMID: 24553167.

- 2. Hammad IA, Chauhan SP, Magann EF, Abuhamad AZ. Peripartum complications with cesarean delivery: a review of Maternal-Fetal Medicine Units Network publications. The journal of maternal-fetal & neonatal medicine: the official journal of the European Association of Perinatal Medicine, the Federation of Asia and Oceania Perinatal Societies, the International Society of Perinatal Obstet. 2014;27(5):463-74. Epub 2013/09/07. doi: 10.3109/14767058.2013.818970. PubMed PMID: 24007280.
- 3. Moshiri M, Osman S, Bhargava P, Maximin S, Robinson TJ, Katz DS. Imaging evaluation of maternal complications associated with repeat cesarean deliveries. Radiologic clinics of North America. 2014;52(5):1117-35. Epub 2014/09/01. doi: 10.1016/j.rcl.2014.05.010. PubMed PMID: 25173662.
- 4. Smaill FM, Grivell RM. Antibiotic prophylaxis versus no prophylaxis for preventing infection after cesarean section. The Cochrane database of systematic reviews. 2014;10:Cd007482. Epub 2014/10/29. doi: 10.1002/14651858.CD007482.pub3. PubMed PMID: 25350672.
- 5. Lyon JB, Richardson AC. Careful surgical technique can reduce infectious morbidity after cesarean section. American journal of obstetrics and gynecology. 1987;157(3):557-62. Epub 1987/09/01. PubMed PMID: 3307420.
- 6. Brocato BE, Thorpe EM, Jr., Gomez LM, Wan JY, Mari G. The effect of cesarean delivery skin incision approach in morbidly obese women on the rate of classical hysterotomy. Journal of pregnancy. 2013;2013:890296. Epub 2013/12/19. doi: 10.1155/2013/890296. PubMed PMID: 24349784; PubMed Central PMCID: PMCPmc3853441.
- 7. Aird LN, Brown CJ. Systematic review and meta-analysis of electrocautery versus scalpel for surgical skin incisions. American journal of surgery. 2012;204(2):216-21. Epub 2012/04/28. doi: 10.1016/j.amjsurg.2011.09.032. PubMed PMID: 22537473.
- 8. Carter PL. The life and legacy of William T. Bovie. American journal of surgery. 2013;205(5):488-91. Epub 2013/04/18. doi: 10.1016/j.amjsurg.2012.12.005. PubMed PMID: 23592153.
- 9. Vender JR, Miller J, Rekito A, McDonnell DE. Effect of hemostasis and electrosurgery on the development and evolution of brain tumor surgery in the late 19th



- and early 20th centuries. Neurosurgical focus. 2005;18(4):e3. Epub 2005/04/23. PubMed PMID: 15844866.
- 10. Johnson CD, Serpell JW. Wound infection after abdominal incision with scalpel or diathermy. The British journal of surgery. 1990;77(6):626-7. Epub 1990/06/01. PubMed PMID: 2143426.
- 11. Ji GW, Wu YZ, Wang X, Pan HX, Li P, Du WY, Qi Z, Huang A, Zhang LW, Zhang L, Chen W, Liu GH, Xu H, Li Q, Yuan AH, He XP, Mei GH. Experimental and clinical study of influence of high-frequency electric surgical knives on healing of abdominal incision. World journal of gastroenterology: WJG. 2006;12(25):4082-5. Epub 2006/07/01. PubMed PMID: 16810765; PubMed Central PMCID: PMCPmc4087727.
- 12. Rappaport WD, Hunter GC, Allen R, Lick S, Halldorsson A, Chvapil T, Holcomb M, Chvapil M. Effect of electrocautery on wound healing in midline laparotomy incisions. American journal of surgery. 1990;160(6):618-20. Epub 1990/12/01. PubMed PMID: 2147542.
- 13. Ly J, Mittal A, Windsor J. Systematic review and meta-analysis of cutting diathermy versus scalpel for skin incision. The British journal of surgery. 2012;99(5):613-20. Epub 2012/03/01. doi: 10.1002/bjs.8708. PubMed PMID: 22367850.
- 14. (NICE). NIfHaCE. Surgical-site Infection. Prevention and Treatment of Surgical-site Infection. NICE Clinical Guideline. NICE. 2008:74.
- 15. Shamim M. Diathermy vs. scalpel skin incisions in general surgery: double-blind, randomized, clinical trial. World journal of surgery. 2009;33(8):1594-9. Epub 2009/05/07. doi: 10.1007/s00268-009-0064-9. PubMed PMID: 19418093.
- 17. Dixon AR, Watkin DF. Electrosurgical skin incision versus conventional scalpel: a prospective trial. Journal of the Royal College of Surgeons of Edinburgh. 1990;35(5):299-301. Epub 1990/10/01. PubMed PMID: 2283608.



Protocol version: 1.0 Page **10** of **11** 

- 18. Elmar A. Joura, M.D., Peter Husslein, M.D. Case Report on Cesarean Delivery, Bladder Flap and use of diathermy. The journal of Reproductive Medicine.
- J Reprod Med 2000;45:363-364.
- 19. Charoenkwan K, Chotirosniramit N, Rerkasem K. Scalpel Versus Elctrosurgery for abominal incisions . Cochrane Database of Systemic Reviews, 2012. CD005987.

Texas Tech University Health Sciences Center IRB NUMBER: L15-144 IRB APPROVAL DATE: 06/17/2015